CLINICAL TRIAL: NCT00532818
Title: Randomized, Double-Blind, Phase III Trial of Chemotherapy Plus the Transcriptional Therapy Hydralazine and Magnesium Valproate Versus Chemotherapy Plus Placebo in Recurrent and Metastatic Cervical Cancer.
Brief Title: Hydralazine Valproate for Cervical Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Institute of Cancerología (Other Government)
Collaborators: Psicofarma, S.A. De C.V. (Industry)
Responsible Party: Lucely Cetina, Instituto Nacional de Cancerologia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 006/027/ICI
Record Dates: First submitted 2007-09-18; First posted 2007-09-20 (Estimated); Last update posted 2009-03-30 (Estimated); Status verified 2009-03

CONDITIONS: Metastatic Cervical Cancer
Keywords: Epigenetic therapy; Hydralazine; Valproate; Cervical cancer; Randomized; Phase III
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Hydralazine; Valproic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator)
  Interventions: Drug: Placebo
- 2 (Experimental)
  Interventions: Drug: Hydralazine and magnesium valproate

INTERVENTIONS:
Drug: Hydralazine and magnesium valproate — Cisplatin + Topotecan plus hydralazine valproate
  Other Names: TRANSKRIP R/L
  Arms: 2
Drug: Placebo — Cisplatin + Topotecan plus placebo
  Other Names: TRANSKRIP R/L
  Arms: 1

SUMMARY:
The current standard for recurrent, persistent or metastatic cervical cancer is palliative chemotherapy with cisplatin topotecan, however, the results need to be improved. Epigenetic aberrations play an important role in cancer progression by silencing growth regulatory genes and there is now evidence that inhibitors of DNA methylation and HDAC inhibition synergize the cytotoxicity of chemotherapy.

Objective. To determine the superiority of epigenetic therapy with hydralazine and valproate plus standard cisplatin topotecan against placebo plus cisplatin topotecan upon progression-free survival.

Hypothesis. Hydralazine and magnesium valproate associated to cisplatin topotecan will increase progression-free survival from 4.6 to 7.6 months as compared with the same regimen of chemotherapy plus placebo.

DETAILED DESCRIPTION:
Randomized, double-blind phase III trial. A total of 143 patients (alpha 0.5, power 0.8)with metastatic, persistent or recurrent cervical cancer without previous systemic treatment will be randomized to cisplatin topotecan + placebo or cisplatin topotecan hydralazine valproate for 6 courses every 3 weeks. Patients will receive an oral dose of hydralazine of 182mg (rapid) or 83mg (slow) according to the acetylator phenotype in a single daily dose and magnesium valproate at an oral dose of 40mg/Kg t.i.d. Both drugs in a slow-release formulation. Experimental drugs or placebo will start from seven days before day 1 of chemotherapy until the end of the sixth course.

ELIGIBILITY:
Inclusion Criteria:

* informed consent, histological diagnosis of persistent, recurrent or metastatic cervical carcinoma; measurable disease by physical examination, CT Scan, MRI or PET-CT. Biopsy is required for confirmation only if the lesion is unique, has less than 2cm in the longest diameter or has no clearly defined borders.
* Patients should have no previous systemic treatment (could have received chemotherapy as radiosensitization to the pelvis and or para-aortic field.
* Aged >18 years, performance status 0-2 according to ECOG classification, and adequate liver, hematological and renal function, as defined by: hemoglobin >10 g/L, leukocytes >4000/mm3, platelets >100 000mm3; normal creatinine value and creatinine clearance >60 mL/min; total bilirubin < 1.5 upper normal limit value.

Exclusion Criteria:

* History of allergy to hydralazine or valproate; past or present condition of rheumatic disease, central nervous system disease, heart failure from aortic stenosis and postural hypotension as diagnosed by a physician; newly diagnosed hypertension patients with or without pharmacological treatment are allowed as long as their treatment do not include hydralazine.
* Previous use of the experimental drugs (hydralazine and magnesium valproate) as well as if patients were pregnant or breast-feeding. Other exclusion criteria are uncontrolled systemic disease or infection.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Estimated)
Dates: Start 2007-07; Primary Completion 2010-09 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 2-years

SECONDARY OUTCOMES:
Response rate, safety, overall survival. | 2-years

CONTACTS AND LOCATIONS:
Overall Officials: Myrna Candelaria, MD, Study Chair — Instituto Nacional de Cancerologia, Columbia
Locations (1):
- Instituto Nacional de Cancerologia, Mexico City, Mexico City, Mexico

REFERENCES:
- See also: Related Info — http://www.incan.org.mx